CLINICAL TRIAL: NCT03942588
Title: High-intensity Interval Training for Adults With Chronic Stroke Impairments: A Pilot Feasibility Study
Brief Title: High-intensity Interval Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Pamela Rogers Bosch, Associate Professor, Northern Arizona University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1002492
Record Dates: First submitted 2019-02-14; First posted 2019-05-08 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Exercise Intervention group and Usual Activity Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Twice-weekly supervised high-intensity interval treadmill training in a laboratory setting for 10 weeks.
  Interventions: Behavioral: High-intensity interval training
- Control (No Intervention): Usual activities for 10 weeks

INTERVENTIONS:
Behavioral: High-intensity interval training
  Arms: High-intensity interval training

SUMMARY:
Aerobic conditioning is very important after stroke as it may reduce the risk of subsequent stroke and overall mortality. High-intensity interval training (HIIT), in which aerobic training workload is varied between lower and higher intensity bouts within a training session, is known to be effective for maximizing aerobic capacity in healthy individuals and those with cardiac disease. HIIT has not been studied extensively in adults with stroke, but it could be an efficient way to maximize aerobic capacity in this population. Furthermore, using heart rate response to establish training intensity may lead to underestimation of target intensity after stroke because blood pressure medications may blunt the heart rate response. Ventilatory threshold is an alternate method of establishing training intensity and is derived independently of heart rate response. The investigators hypothesized that a 10-week program of treadmill HIIT with intensity based on ventilatory threshold would be feasible in adults at least 6 months post-stroke, and would increase aerobic capacity.

DETAILED DESCRIPTION:
Stroke is the main cause of serious, long-term disability among Americans. The effects of a stroke make it difficult to participate in routine, daily activities so people become seriously deconditioned after a stroke. This increases the chances of having another stroke and it also increases the risk of death. Even a small increase in aerobic capacity reduces these risks, making aerobic training an important component of post-stroke management.

Twenty to 60 minutes of moderate-intensity exercise on most days of the week is recommended for people with cardiovascular disease, but this is not very practical for many people after a stroke, who need to practice functional tasks like using the impaired arm and improving walking and balance. Another problem is that even when people do participate in aerobic training after a stroke, the improvements in aerobic capacity are sometimes surprisingly small. It is possible that the intensity of the training program was inadequate to improve aerobic capacity in some interventions. High-intensity interval training, in which people alternate between short, intense bouts of exercise and recovery bouts within the session, may be a way to improve aerobic capacity after a stroke with a more feasible training schedule that leaves time to practice functional skills too. High-intensity interval training on a treadmill might be appropriate to improve aerobic capacity and walking ability.

This non-randomized, non-blinded pilot study was designed to assess the feasibility of ten weeks of high-intensity interval training (HIIT) using treadmill training for adults with impaired walking who were at least 6 months post-stroke.

A secondary objective was to measure change in aerobic capacity, and a tertiary objective was to measure functional change in self-selected walking speed and leg strength as a result of the intervention.

10 participants completed HIIT intervention while 5 participants served as controls and received no intervention, but completed both baseline and post-testing sessions.

HIIT participants completed twice-weekly, 35-minute training sessions in a research laboratory for 10 consecutive weeks. At baseline and 12 weeks, all participants completed a graded exercise test, 10-meter walk test at self-selected and fastest, safe overground walking speeds, and a 30-second sit-to-stand test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18 years of age or older who had a unilateral stroke at least 6 months prior to enrollment
* Ability to provide informed consent and follow instructions to participate
* Medically stable
* Must be able to walk with no more than contact guard assistance on level surfaces
* Must be willing to walk on a treadmill with a support harness and handrail

Exclusion Criteria:

* Cerebellar stroke
* Medical instability
* Implanted pacemaker or defibrillator
* Inability to walk on a treadmill with a support harness and use of handrail for at least 5 minutes
* Absence of walking impairments
* Abnormal resting heart rate, blood pressure or ECG
* Abnormal ECG during graded exercise test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic Capacity | Baseline and 12 weeks
  Whole-body oxygen consumption measured via a graded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Pamela R Bosch, PhD, Principal Investigator — Northern Arizona University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosch PR, Holzapfel S, Traustadottir T. Feasibility of Measuring Ventilatory Threshold in Adults With Stroke-Induced Hemiparesis: Implications for Exercise Prescription. Arch Phys Med Rehabil. 2015 Oct;96(10):1779-84. doi: 10.1016/j.apmr.2015.04.023. Epub 2015 May 12. PMID 25979162
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Tang A, Marzolini S, Oh P, McIlroy WE, Brooks D. Factors associated with change in aerobic capacity following an exercise program for individuals with stroke. J Rehabil Med. 2013 Jan;45(1):32-7. doi: 10.2340/16501977-1053. PMID 23150062
- [Background] Moholdt TT, Amundsen BH, Rustad LA, Wahba A, Lovo KT, Gullikstad LR, Bye A, Skogvoll E, Wisloff U, Slordahl SA. Aerobic interval training versus continuous moderate exercise after coronary artery bypass surgery: a randomized study of cardiovascular effects and quality of life. Am Heart J. 2009 Dec;158(6):1031-7. doi: 10.1016/j.ahj.2009.10.003. PMID 19958872
- [Background] Calmels P, Degache F, Courbon A, Roche F, Ramas J, Fayolle-Minon I, Devillard X. The feasibility and the effects of cycloergometer interval-training on aerobic capacity and walking performance after stroke. Preliminary study. Ann Phys Rehabil Med. 2011 Feb;54(1):3-15. doi: 10.1016/j.rehab.2010.09.009. Epub 2010 Nov 18. English, French. PMID 21131249
- See also: Conference Abstract — https://doi.org/10.1016/j.apmr.2017.08.022